CLINICAL TRIAL: NCT01628185
Title: Pain Assessment in the Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 11-0691
Record Dates: First submitted 2012-02-23; First posted 2012-06-26 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Delirium; Critical Illness
MeSH Terms: conditions — Delirium; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pain Observations: Adult ICU patients who are not comatose with Richmond Agitation-Sedation Scale (RASS) score of -3 to 4 and unable to self-report pain. Patients will be excluded for neurological deficits (acute or chronic) that prevent observation of the muscle tonus or movement
  Interventions: Procedure: Repositioning

INTERVENTIONS:
Procedure: Repositioning — pain assessment at baseline then following routine care repositioning in bed

SUMMARY:
Pain assessment using self-report scales (Visual Analogue Scale, Numerical Rating Scale), is recommended in the general population, however it is not always possible in patients with altered neurological status such as sedated patients or patients with delirium. Consequently, pain assessment is highly challenging in these ICU patients. This is a prospective observational study assessing 3 behavioral pain scales in the ICU.

The hypothesis of this proposal is that one of the three ICU pain scales has a more important reliability than the others. Such a scale could be recommended to be used to measure pain intensity in ICU patients not able to communicate.

DETAILED DESCRIPTION:
The aims of this observational study are to measure and compare the psychometric properties of Behavioral Pain Scale (BPS), Critical Care Pain Observation Tool (CPOT) and Non Verbal Pain Scale (NVPS) at baseline and following repositioning procedure in the ICU

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* not comatose, defined by a Richmond Agitation Sedation Scale (RASS) ≥ -3, i.e. between -3 and +4
* not able to self-report accurately their pain intensity using a visually enlarged 0-10 numeric rating scale

Exclusion Criteria:

-neurological deficits (acute or chronic) that prevent observation of the muscle tonus or movement. For example:

* Quadriplegia
* Current use of Neuromuscular blocking agents
* Severe brain injuries

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensive Care Unit patients
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
pain score reliability | change from time 0 pain assessment to time 30min pain assessment
  Behavioral Pain Scale(BPS), Critical Care Pain Observation Tool (CPOT), Non Verbal Pain Scale (NVPS)

SECONDARY OUTCOMES:
pain score validity | change from time 0 pain assessment to time 30min pain assessment
  Behavioral Pain Scale(BPS), Critical Care Pain Observation Tool (CPOT), Non Verbal Pain Scale (NVPS)

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Hall, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Chanques G, Pohlman A, Kress JP, Molinari N, de Jong A, Jaber S, Hall JB. Psychometric comparison of three behavioural scales for the assessment of pain in critically ill patients unable to self-report. Crit Care. 2014 Jul 25;18(5):R160. doi: 10.1186/cc14000. PMID 25063269